CLINICAL TRIAL: NCT01915667
Title: Bioavailability Study Comparing Two Solid Oral Formulations of GLPG0634 in Healthy Male Subjects
Brief Title: Oral Bioavailability of Two Solid Formulations of GLPG0634
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLPG0634-CL-107
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG0634; Capsules; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GLPG0634 capsule fasted (Experimental): Single dose of GLPG0634 as capsules in fasted condition
  Interventions: Drug: 200 mg GLPG0634 as capsules, fasted
- GLPG0634 tablet fasted (Experimental): Single dose of GLPG0634 as tablets in fasted condition
  Interventions: Drug: 200 mg GLPG0634 as tablets, fasted
- GLPG0634 tablet fed (Active Comparator): Single dose of GLPG0634 as tablets in fed condition
  Interventions: Drug: 200 mg GLPG0634 as tablets, fed

INTERVENTIONS:
Drug: 200 mg GLPG0634 as capsules, fasted — single oral dose of 200 mg GLPG0634 given as capsules in fasted condition
  Arms: GLPG0634 capsule fasted
Drug: 200 mg GLPG0634 as tablets, fasted — single oral dose of 200 mg GLPG0634 given as tablets in fasted condition
  Arms: GLPG0634 tablet fasted
Drug: 200 mg GLPG0634 as tablets, fed — single oral dose of 200 mg GLPG0634 given as tablets in fed condition
  Arms: GLPG0634 tablet fed

SUMMARY:
The purpose of the study is to evaluate the amount of compound present in the blood (relative bioavailability) after a single administration of GLPG0634 as a tablet versus a capsule in fasted conditions in male healthy subjects.

Also, the effect of food on the bioavailability of the tablet formulation will be studied as well as the safety and tolerability of single oral doses of GLPG0634 given either as capsule or tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, age 40-60 years
* BMI between 18-30 kg/m2

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The amount of GLPG0634 and metabolite in plasma after a single dose of GLPG0634 as capsules or tablets | From predose (before first study drug administration) up to 144 hours post last study drug administration
  To characterize and compare the amount of GLPG0634 and metabolite in plasma (relative bioavailability) in male healthy subjects after a single administration of either a capsule or tablet formulation in a fasted condition. For the tablet formulation, also the amount of GLPG0634 and metabolite in plasma will be evaluated after fasting and in fed condition.

SECONDARY OUTCOMES:
The number of subjects with adverse events, abnormal lab tests, physical examinations, vital signs and ECG after a single dose of GLPG0634 as capsules or tablets | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG0634 after a single oral dose as capsules or tablets, either fasted or fed, in male healthy subjects in terms of adverse events (AEs), abnormalities in laboratory tests, physical examinations, vital signs and electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Pille Harrison, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Antwerp, Belgium